CLINICAL TRIAL: NCT01934088
Title: Nurse Administered Propofol Sedation vs. Standard Therapy for Colonoscopy in Patients With IBD. A Randomised Controlled Study on Satisfaction and Adherence to Treatment Program.
Brief Title: Satisfaction With Nurse Administered Propofol Sedation vs. Midazolam With Fentanyl Sedation for Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Jeppe Thue Jensen, MD, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013052044 v.1
Record Dates: First submitted 2013-08-12; First posted 2013-09-04 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Inflammatory Bowel Disease; Endoscopy; Sedation
Keywords: Inflammatory Bowel disease; IBD; Sedation; NAPS; Propofol; Midazolam; Satisfaction; Feasibility
MeSH Terms: conditions — Inflammatory Bowel Diseases; Personal Satisfaction | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Experimental): Propofol in refract doses. Induction: 10-60 mg supplemented with 10-30 mg following an age correlated algorithm. Maintenance with refract bolus of 10-20 mg every 1-2 minutes after assessed need and condition
  Interventions: Drug: Propofol
- Fentanyl and Midazolam (Active Comparator): 0.025-0.05 mg of Fentanyl i.v. minimum 5 minutes before procedure as a single shot. Midazolam 1-2 mg i.v. for induction and 0.5-1 mg i.v. for maintenance after assessing needs and condition
  Interventions: Drug: Midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol
  Arms: Propofol
Drug: Midazolam
  Other Names: Midazolam "Hameln" ATC-code: N05CD08
  Arms: Fentanyl and Midazolam
Drug: Fentanyl
  Other Names: Fentanyl "Hameln" ATC-code: N01AH01
  Arms: Fentanyl and Midazolam

SUMMARY:
Sedation for endoscopy is a service more than a necessity. Therefore it should be patient driven. Patients with inflammatory bowel disease (IBD) undergoes life long endoscopic control. Therefore, satisfaction with the procedure experience is paramount for patients with IBD. Investigators wish to study the feasibility and the effect on patient experience of two drugs. Propofol administered by endoscopy nurses (NAPS) and conventional therapy with a combination of fentanyl and midazolam. Investigators hypothesize that patients sedated with propofol has a better procedure experience, that a well performed sedation equals a better experience and that NAPS is as feasible as fentanyl with midazolam sedation.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory Bowel Disease (IBD) or suspected IBD
* Planned Endoscopy
* Candidate for propofol sedation
* willingness to be randomized
* Ability to complete questionnaire

Exclusion Criteria:

* Allergy to drugs
* American Society of Anesthesiologists Class III
* Body Mass Index > 35
* Ventricular retention
* Acute condition
* Severe Chronic obstructive pulmonary disease
* Sleep apnea
* Potentially difficult airway or previous difficulty with anesthesia
* Pregnancy
* <18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Satisfaction | Participants will be interviewed when an Aldrete recovery score of 12 is achieved, an expected average of 2 hours after admission
  Satisfaction points in a post procedure questionnaire.

SECONDARY OUTCOMES:
Pre-disposing factors for satisfaction with procedure and sedation | At admission to the hospital at time 0
  pre-operative questionnaire

OTHER OUTCOMES:
Correlation between quality of sedation and satisfaction | At the end of procedure, an expected average of 1 hour after admission
  Sedation efficacy is measured through use of a previously developed competency assessment tool. The quality of sedation score. The score is correlated with patient satisfaction
Feasibilty of method | participants will be followed for the duration of hospital stay, an expected average of 2 hours
  Timespand from entering the OR until discharge. Safety parameters during sedation. Number of adverse events, number of airway interventions, number of rescue treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Thue Jensen, MD, Principal Investigator — Gastroenheden D, endoscopy, Herlev Hospital; Peter Vilmann, Professor, Study Director — Gastroenheden D, Endoscopy, Herlev Hospital
Locations (1):
- Endoscopy, Gastrounit, Herlev Hospital, Herlev, Region H, Denmark

REFERENCES:
- [Background] Jensen JT, Vilmann P, Horsted T, Hornslet P, Bodtger U, Banning A, Hammering A. Nurse-administered propofol sedation for endoscopy: a risk analysis during an implementation phase. Endoscopy. 2011 Aug;43(8):716-22. doi: 10.1055/s-0030-1256515. Epub 2011 Aug 2. PMID 21811940
- [Derived] Steenholdt C, Jensen JT, Brynskov J, Moller AM, Limschou AC, Konge L, Vilmann P. Patient Satisfaction of Propofol Versus Midazolam and Fentanyl Sedation During Colonoscopy in Inflammatory Bowel Disease. Clin Gastroenterol Hepatol. 2022 Mar;20(3):559-568.e5. doi: 10.1016/j.cgh.2020.10.037. Epub 2020 Oct 22. PMID 33371995